CLINICAL TRIAL: NCT03850288
Title: Inhibitory Control in Eating Disorders (Anorexia Nervosa, Bulimia Nervosa and Binge Eating Disorder)
Brief Title: Inhibitory Control and Eating Disorders
Acronym: InhibEating
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0621
Record Dates: First submitted 2019-02-15; First posted 2019-02-21 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-01

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa; Binge Eating
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Bulimia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anorexia Nervosa: Patients with a diagnosis of anorexia nervosa (According to the DSM-V criteria). These patients are characterized by a restriction of food intake leading to weight loss or a failure to gain weight resulting in a "significantly low body weight" of what would be expected for someone's age, sex and height. Moreover, there is a fear of becoming fat or of gaining weight.Then, these patients have a distorted view of themselves and of their condition.
  Interventions: Other: Neuropsychological assessment : Stroop task; Other: Neuropsychological assessment : Go No Go task
- Bulimia Nervosa: Patients with a diagnosis of bulimia nervosa. According to the DSM-V criteria, these patients are characterized by recurrent episodes of binge eating (eating, in a discrete period of time, an amount of food that is definitely larger than most people would eat during a similar period of time and under similar circumstances), a sense of lack of control over eating during the episode, recurrent inappropriate compensatory behaviour in order to prevent weight gain, such as self-induced vomiting, misuse of laxatives, diuretics, or other medications, fasting, or excessive exercise.
  The binge eating and inappropriate compensatory behaviours both occur, on average, at least once a week for three months. Moreover, there is a self-evaluation influenced by body shape and weight.
  Interventions: Other: Neuropsychological assessment : Stroop task; Other: Neuropsychological assessment : Go No Go task
- Binge Eating Disorder: Patients with a diagnosis of Binge Eating Disorder. These patients are characterized by recurrent episodes of binge eating (eating, in a discrete period of time (e.g. within any 2-hour period), an amount of food that is definitely larger than most people would eat during a similar period of time and under similar circumstances), a sense of lack of control over eating during the episode. The binge eating episodes are associated with three or more of the following: eating much more rapidly than normal, eating until feeling uncomfortably full, eating large amounts of food when not feeling physically hungry, eating alone because of feeling embarrassed by how much one is eating, feeling disgusted with oneself, depressed or very guilty afterward,marked distress regarding binge eating is present. Moreover, binge eating occurs, on average, at least once a week for three months
  Interventions: Other: Neuropsychological assessment : Stroop task; Other: Neuropsychological assessment : Go No Go task

INTERVENTIONS:
Other: Neuropsychological assessment : Stroop task — Stroop task is an interference task assessing cognitive inhibitory control. This "paper-and-pencil" task aims to evaluate the inhibition of an automated process such as reading by asking participants to name the color of color names written in a different color ink.
  This test is non-invasive.
Other: Neuropsychological assessment : Go No Go task — Go No Go task assessing motor inhibitory control. This computer-based task is designed to evaluate motor inhibition by asking participants to respond to a stimulus as quickly as possible by inhibiting another distractor stimulus.
  This test is non-invasive.

SUMMARY:
Executive functions are part of the high-level cognitive processes essential to the proper functioning of human cognition. They consist mainly of flexibility, updating and inhibition. Some studies have shown a correlation between executive disorders (impaired executive function) and psychiatric disorders such as obsessive-compulsive disorder or phobias. These executive disorders are related to dysfunctions of the fronto-striatal loops.

In addition, other studies have investigated the link that may exist between eating disorders such as anorexia or bulimia nervosa and executive functioning. Anorexia nervosa, bulimia nervosa and binge eating disorders are eating disorders characterized by a dysfunction in food intake with restriction of food or compulsions as well as strong concerns about the body schema. Concerning the executive functioning, these studies highlight a lack of cognitive flexibility for patients with anorexia nervosa and bulimia nervosa but also dysfunctions depending on the type of pathology (anorexia nervosa or bulimia nervosa). These studies also highlight the beneficial effects of cognitive remediation on people with eating disorders.

However, the investigation of the inhibitory control has not yet been specifically studied. Moreover, since eating disorders are structurally different, a comparison between several pathologies would be interesting to consider.

The aim of this study is to determine if a dysfunction of inhibitory control can be highlighted in people with eating disorders. This study would also allow further researches about cognitive remediation suitable for the specific difficulties encountered in these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 19 to 40 years old
* Patient with a BMI between 13 and 40 kg/m2
* Outpatients of the Refering Center of Eating Disorders ('Hospices Civils de Lyon' in Lyon) suffering of an eating disorder diagnosis (Anorexia Nervosa, Bulimia Nervosa or Binge Eating Disorder)
* Patient who agrees to participate to the study.

Exclusion Criteria:

* Patient with psychiatric comorbidity severe (DSM V) and not stable (during the 8 weeks before inclusion)
* Patient with psychotropic treatment (started or modified during the 8 weeks before inclusion)
* Major patient protected by a measure of legal protection
* Patient younger than 19 years old
* Participation to another study at the same time

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women aged 19 to 40 years old, with a BMI between 13 and 40 kg/m2, outpatients of the Refering Center of Eating Disorders ('Hospices Civils de Lyon' in Lyon), with an eating disorder diagnosis (Anorexia Nervosa, Bulimia Nervosa or Binge Eating Disorder).
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Inhibition processes assessment - the Stroop task, Execution time | 1 day
  Execution time in the Stroop task
Inhibition processes assessment - the Stroop task, Errors | 1 day
  Errors in the Stroop task
Inhibition processes assessment - the Go No Go task, Execution time | 1 day
  Execution time in the Go No Go task.
Inhibition processes assessment - the Go No Go task, Variability of execution time | 1 day
  Variability of execution time in the Go No Go task
Inhibition processes assessment - the Go No Go task, Errors | 1 day
  Errors in the Go No Go task

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Référent pour l'Anorexie et les Troubles du Comportement Alimentaire, Bron, France

IPD SHARING:
Plan to Share IPD: No